CLINICAL TRIAL: NCT04090008
Title: A Randomized Controlled Trial on Platelet Rich Plasma Gel Compared to Normal Saline Dressing of Diabetic Foot Ulcers
Brief Title: A Randomized Trial on Platelet Rich Plasma Versus Saline Dressing of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mansoura103
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP gel (Active Comparator): PRP gel was applied to the ulcer twice per week after preparation and then the ulcer was covered with Vaseline gauze, few layers of sterile gauze and crepe bandage.
  Interventions: Drug: PRP gel
- Saline dressing (Active Comparator): daily dressing of the ulcer with normal saline was done
  Interventions: Drug: Saline dressing

INTERVENTIONS:
Drug: PRP gel — The PRP gel is applied on the ulcer twice per week
  Arms: PRP gel
Drug: Saline dressing — Normal saline is used for dressing of the ulcer twice a week
  Arms: Saline dressing

SUMMARY:
New treatments for persistent DFU have emerged, among which are the bioengineered skin substitutes, extracellular matrix proteins products, matrix metalloproteinases modulators, and growth factor therapy. Platelet rich plasma (PRP) gel has been used for stimulating wound healing since the last decade of the 20th century. This randomized trial was conducted to assess the role of PRP in gel form as a treatment for clean non-healing diabetic foot ulcer in comparison to regular dressing with saline as a control.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of both sexes aging below 70 years with non-infected chronic foot ulcer confined to one anatomical site. Chronicity was defined as non-healing ulcer for twelve or more weeks

Exclusion Criteria:

* Patients with chronic limb ischemia.
* Evidence of osteomyelitis in the affected foot
* Exposed tendons, ligaments or bones at the base of ulcer
* Patients who received radiotherapy or chemotherapy at time of study or within 3 months of its beginning.
* Patients having low peripheral platelet count, low serum albumin level or low hemoglobin level

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the ulcer size | 20 weeks
  the difference between ulcer size before and after treatment subdivided by the ulcer size before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided